CLINICAL TRIAL: NCT07378787
Title: The Effect of Time-Restricted Eating in Combination With a Low Glycaemic Index Diet on Cognitive Function, Markers of Biological Age and Metabolic Health in Late-Perimenopausal and Menopausal Women: a Randomized Controlled Trial. The NutriAge Trial.
Brief Title: Time-Restricted Eating in Combination With a Low Glycaemic Index Diet on Cognitive Function, Biological Ageing and Metabolic Health in Perimenopause and Menopause.
Acronym: NutriAge
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nicosia (Other)
Collaborators: Digital Diet Clinic Ltd (Unknown); GENOS LIMITED (Unknown)
Responsible Party: Principal Investigator, Elena Philippou, Associate Professor Nutrition-Dietetics, University of Nicosia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EEBK/EΠ/2025/52
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Late-perimenopause; Menopause; Perimenopause
Keywords: Peri-menopause; menopause; intermittent fasting; low glycaemic-index diet; women; time-restricted eating; biological ageing; metabolic markers; cognitive function; cognition; tender joints; swollen joints; nutrition; microbiome; Mediterranean diet; GlycanAge; randomized controlled trial; BDNF; insulin resistance; middle-aged; global health
MeSH Terms: conditions — Intermittent Fasting; Insulin Resistance | interventions — Diet, Mediterranean

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time-Restricted Low Glycaemic Index Diet (Experimental): Participants in the Time-Restricted-Low-Glycaemic Index group will follow a 16:8 intermittent fasting regimen, where all meals are consumed within an 8-hour eating window. Their diet will also consist of low-glycaemic index foods following the principles of the Mediterranean diet. They will provided with individualized dietary plans through the Nutrium App and followed up regularly through the app.
  Interventions: Other: Time-Restricted Low-Glycaemic Index Diet
- Control group (No Intervention): The Control Group will receive no dietary intervention during the 6-month trial but will be placed on a waiting list for future guidance if requested. Their dietary intake will be recorded through the Nutrium App.

INTERVENTIONS:
Other: Time-Restricted Low-Glycaemic Index Diet — The combination of a 16:8 Time-Restricted eating period with a low glycaemic index Mediterranean diet
  Other Names: intermittent fasting; low glycaemic diet; Mediterranean diet; 16:8
  Arms: Time-Restricted Low Glycaemic Index Diet

SUMMARY:
The goal of this randomised controlled trial is to investigate whether Time-Restricted Eating (TRE) combined with a Low Glycaemic Index Mediterranean Diet can improve cognitive function, metabolic health, and biological ageing in late perimenopausal and menopausal women aged 45-75 years with a BMI ≥23 kg/m². It will consist of a 12-week intervention followed by a 12 week follow-up period.

Researchers will compare a group following the 16:8 time-restricted eating schedule and Low Glycaemic Index Mediterranean Diet to a control group (waiting list) receiving no dietary or meal-timing instructions to determine if these dietary strategies influence cognitive function, assessed via brain-derived neurotropic factor (BDNF) and cognitive function tests, metabolic outcomes, biological age, the gut microbiome, tender and swollen joint count and global health.

Participants will:

Follow a 16:8 time-restricted eating schedule (eating within an 8-hour window and fasting for 16 hours) if assigned to the intervention group.

Adhere to a tailored Low Glycaemic Index Mediterranean Diet and track meals using the Nutrium app.

Attend study visits at the University of Nicosia at Week 0, Week 12, and Week 24 for various assessments.

Provide biological samples, including blood samples at five specific intervals and stool samples at Week 0 and Week 12.

Complete multiple questionnaires regarding diet, lifestyle, sleep quality, physical activity, tender and swollen joints, and quality of life.

Undergo physical and cognitive assessments, such as CNS Vital Signs tests, blood pressure measurements, and body composition analysis.

The two groups will be compared to understand if the intervention improves outcomes and can thus be applied in this population group.

DETAILED DESCRIPTION:
This randomized controlled trial will run over a period of 24 weeks (6 months) and will be divided into two main phases: a 12-week intervention phase followed by a 12- week follow-up phase designed to assess long-term adherence and health outcomes. The participants will be randomized to one of two groups: the intervention group of a Time-Restricted Eating combined with a Low Glycaemic Index diet (TRE-LGI) group, and the control group which will not receive any dietary intervention.

During the intervention phase (Week 0 to Week 12), participants randomized to the TRE-LGI group will follow a structured eating plan. They will be instructed to consume all their meals within an 8-hour eating window each day and adhere to a low glycaemic index Mediterranean-style diet. Participants randomized to the control group will not receive any dietary intervention but will continue to be monitored for study purposes.

Assessments will be conducted at three time points during this phase. At baseline (Week 0), participants will complete a full set of evaluations, including the online Computerised Neurocognitive Testing tool CNS Vital Signs, metabolic markers (insulin sensitivity, and lipid profiles, C-reactive protein (CRP), BDNF assessment using Enzyme-Linked Immunosorbent Assay (ELISA) Test, biological ageing assessment using the N-glycome analysis (GlycanAge test), gut microbiome analysis from stool samples, body composition, blood pressure, waist circumference, sleep quality using the Pittsburgh Sleep Quality Index (PSQI), physical activity using the International Physical Activity Questionnaire-Short Form IPAQ-SF, tender and swollen joint count and Global Health using the PROMIS® Scale v1.2 - Global Health.

At Week 6, only the N-glycome composition analysis (GlycanAge) will be repeated to monitor changes in biological ageing.

At Week 12, all baseline assessments will be repeated to measure the effects of the intervention.

The follow-up phase, spanning from week 12-24, will focus on evaluating the participants' ability to sustain the dietary practices achieved during the intervention period without receiving further active dietary guidance. Monitoring will continue to measure the longer-term effects on cognitive, metabolic, and biological health outcomes.

At Week 18, participants will undergo N-glycome composition analysis (GlycanAge) to continue monitoring biological ageing.

At Week 24, a final comprehensive assessment will be conducted, including cognitive function (CNS Vital Signs), BDNF Test, N-glycome analysis, body composition using BIA, BMI, blood pressure, waist circumference, and sleep quality (PSQI), physical activity (IPAQ-SF), tender and swollen joint count, and Global Health PROMIS questionnaire.

Participants in the control group will complete the same assessments at each scheduled time point, allowing for direct comparisons; however, they will not undergo any dietary intervention throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Women in late perimenopausal or menopausal status Note: Late perimenopause is defined as two or more skipped cycles and at least 60 days of amenorrhea. Recent blood tests showing elevated FSH levels support eligibility for late perimenopause. Menopause is defined as 12 consecutive months without a menstrual cycle.
* BMI ≥23 kg/m2
* Age 45-75 years old
* If using any medication, the dose should be stable for the previous 12 months
* Able to use technology and follow the dietary plan

Exclusion Criteria:

* Diagnosis of mild cognitive impairment (MCI) or Alzheimer's disease (AD). Note: (Self-reported memory complaints are allowed).

  * On hormone replacement therapy (HRT)
  * Medical conditions that significantly affect cognitive or metabolic function including diagnosis of type 1 diabetes, severe metabolic disorders, cardiovascular disease, or neurodegenerative conditions, diagnosed eating disorders or severe mental health conditions.
  * Currently enrolled in another intervention.
  * Severe food allergies or dietary restrictions that would prevent adherence to the study diet.
  * History of substance abuse.

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 72 (Estimated)
Dates: Start 2026-01-17 (Actual); Primary Completion 2029-01-20 (Estimated); Study Completion 2029-01-20 (Estimated)

PRIMARY OUTCOMES:
Brain-derived neurotrophic factor concentration | Week 0 and Week 12 for the intervention period and Week 24 for the follow-up period
  Changes between the intervention and control group in the concentration of brain-derived neurotrophic factor assessed by Enzyme-linked Immunosorbent Assay

SECONDARY OUTCOMES:
Cognitive function | Week 0 and Week 12 for the intervention period and Week 24 for the follow-up period
  Cognitive function using CNS Vital Signs assessments, including visual, verbal and composite memory, reaction time, executive function, complex attention and cognitive flexibility
Insulin resistance | Week 0 and Week 12 for the intervention period
  Fasting glucose and insulin to assess insulin resistance using the Homeostatic Model Assessment for Insulin Resistance (HOMA-IR).
Lipid profile | Week 0 and Week 12 for the intervention period
  Total cholesterol, LDL and HDL cholesterol, Triglyceride concentration, the triglyceride-to-HDL (TG/HDL) ratio will be calculated as a predictive marker for cardiovascular risk
C-reactive protein (CRP) | Week 0 and Week 12 for the intervention period
  CRP concentration to assess inflammation
IgG N-glycome composition analysis to assess GlycanAge | The test will be conducted at Week 0, 6, 12, 18, and 24 to monitor progressive changes in biological ageing throughout the 6-month study period.
  The IgG N-glycome composition analysis will be used to measure biological ageing and systemic inflammation by analysing glycans attached to immunoglobulin G (IgG) antibodies in participants' blood samples using high-performance liquid chromatography (HPLC).
Anthropometric measurements: Body weight, height, and calculation of the Body Mass Index | Week 0 and weekly thereafter until Week 24 for body weight and BMI, Week 0: Body height
  Body weight will be measured using minimal clothing. Height will be measured using a standard stadiometer. BMI will be calculated as weight in kg divided by height in metres squared
Body composition analysis using Bioelectrical Impedance Analysis | Week 0 and Week 12 for the intervention phase and Week 24 for the follow-up phase
  Body composition analysis using Bioelectrical Impedance Analysis in the fasted state to assess % body fat, body fat mass, fat-free mass, skeletal muscle mass and visceral fat
Gut microbiome | Week 0 and Week 12 for the intervention period
  Gut microbiome will be assessed by performing phyla-level PCR analysis on the stool sample
Blood pressure | Week 0 and Week 12 of the intervention period and Week 24 of the follow-up period
  Blood pressure will be assessed using standard methods
Sleep duration and quality | Week 0 and Week 12 for the intervention period and Week 24 for the follow-up period
  Subjective assessment of sleep duration and quality using the Pittsburgh Sleep Quality Index (PSQI)
Tender and swollen joint count | Week 0 and Week 12 for the intervention period and Week 24 for the follow-up period
  The participant's number of tender and swollen joints will be self-assessed by providing a diagram to the participant, where they can mark any tender and/or swollen joints.
Global Health | Week 0 and Week 12 for the intervention period and Week 24 for the follow-up period
  Global Health will be assessed using the PROMIS® Scale v1.2 - Global Health which evaluates key domains including global physical health, global mental health, physical function, fatigue, pain interference, emotional distress, social health, and quality of life through Likert-scale items.

OTHER OUTCOMES:
Physical activity assessment | Week 0 and Week 12 for the intervention period and Week 24 for the follow-up period
  Assessment of physical activity will be done using the Physical Activity Questionnaire - Short Form (IPAQ-SF) (confounding outcome)
Nutritional Assessment and adherence to the dietary intervention | Intervention group: weekly monitoring between Week 1 to Week 12. Control group: 3-day food diary at week 1, week 6 and Week 12. All participants: 3-day food diary at Week 18 and Week 24. Adherence to the intervention: week 1, 6, 12, 24
  Energy, macronutrient intake, dietary glycaemic index and timing of eating will be assessed via the Nutrium application. Adherence to the intervention will be assessed via 3-5 day food diaries through the Nutrium app.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Philippou, PhD, Principal Investigator — University of Nicosia
Locations (2):
- Genos Ltd, Zagreb, Croatia
- University of Nicosia, Nicosia, Engomi, Cyprus

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying the results reported in the published article (including cognitive test scores, metabolic markers, and N-glycome markers) will be made available to qualified researchers. Data will be shared only after a formal request and upon approval of a methodologically sound research proposal. To protect participant privacy in accordance with GDPR and the Cyprus National Bioethics Committee, all shared data will be coded, and researchers must sign a Data Use Agreement (DUA) ensuring they will not attempt to re-identify any individual.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available beginning 6 months after the publication of the primary manuscript and ending 10 years after the study start date.
Access Criteria: De-identified individual participant data (IPD) and supporting documents (Study Protocol and SAP) will be made available to qualified academic researchers upon request. To gain access, researchers must submit a detailed research proposal and a methodologically sound analysis plan for review by the NutriAge trial steering committee. Approval is contingent on the scientific merit of the proposal and the feasibility of the analysis. Before data transfer, the requesting institution must execute a Data Use Agreement (DUA) to ensure strict adherence to GDPR standards and to prevent any attempts at participant re-identification.

REFERENCES:
- [Background] Demetriou CA, Hileti D, Onisiphorou E, Kazafanioti C, Alogakos M, Vardakastani D, Christofidou E, Andreou EP, Giannaki CD, Stavrinou PS, Philippou P, Constantinidou F, Philippou E. Associations Between Chrono-Nutrition Behaviours and Cognitive Function in Middle-Aged Adults: The NUTRICO Cross-Sectional Cohort Study. Nutr Bull. 2025 Jun;50(2):262-277. doi: 10.1111/nbu.70000. Epub 2025 Feb 24. PMID 39992029
- See also: Facebook page providing information on study recruitment and progress — https://www.facebook.com/profile.php?id=61582079982648